CLINICAL TRIAL: NCT04524052
Title: Phase I Study to Evaluate the Safety, Tolerability, Pharmacodynamics (PD) and Pharmacokinetics (PK) of DWRX2003 (Niclosamide IM Depot) Injection Following Intramuscular Administration in Healthy Volunteers
Brief Title: To Evaluate Safety, Tolerability, Pharmacodynamics, and Pharmacokinetics of DWRX2003 Against COVID-19
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Daewoong Pharmaceutical Co. LTD. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DWJ1516101_India
Record Dates: First submitted 2020-08-19; First posted 2020-08-24 (Actual); Last update posted 2020-08-24 (Actual); Status verified 2020-08

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- cohort 1 (144 mg) (Experimental): Arms (both) 0.1 mL/site*2 sites Hips (both) 0.2 mL/site*2 sites
  Interventions: Drug: DWRX2003; Drug: Placebo
- cohort 2 (432 mg) (Experimental): Arms (both) 0.3 mL/site *2 sites Hips (both) 0.6 mL/site*2 sites
  Interventions: Drug: DWRX2003; Drug: Placebo
- cohort 3 (960 mg) (Experimental): Arms (both) 0.8 mL/site*2 sites Hips (both) 1.2 mL/site*2 sites
  Interventions: Drug: DWRX2003; Drug: Placebo
- cohort 4 (1200 mg) (Experimental): Arms (both) 1.0 mL/site *2 sites Hips (both) 1.5 mL/site*2 sites
  Interventions: Drug: DWRX2003; Drug: Placebo

INTERVENTIONS:
Drug: DWRX2003 — Intramuscularly injection at pre-defined injection sites
Drug: Placebo — Intramuscularly injection at pre-defined injection sites

SUMMARY:
This study is to assess the safety, tolerability, pharmacodynamics, and pharmacokinetics of Niclosamide (DWRX2003) following escalating doses of DWRX2003 administered as an intramuscular injection in healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

1. Normal healthy human adult male and female volunteers between 18-45 years (both ages inclusive) of age.
2. Volunteers who agree to give written informed consent and are willing to participate in the study.
3. Volunteer having bodyweight minimum of 50 kg.
4. Volunteer having Body Mass Index of 18.50 to 29.90 Kg/m2 (both inclusive).

Exclusion Criteria:

1. Known allergic to Niclosamide or any component of the formulation and to any other related drug.
2. History or presence of significant cardiovascular, respiratory, hepatic, renal, hematological, gastrointestinal, endocrine, immunologic, dermatologic, neurological or psychiatric disease.
3. Female volunteers who are nursing mothers/lactating women or are found positive in beta hCG test.
4. History/ current use of Alcohol or drug abuse.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Estimated)
Dates: Start 2020-08 (Estimated); Primary Completion 2020-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events | follow-up 48 days after dosing
  AE rate, incidence, severity and causality of adverse events (AEs) and serious adverse events (SAEs)

SECONDARY OUTCOMES:
pharmacokinetic changes of niclosamide from baseline in each dose group: Cmax | follow-up 48 days after dosing
  Maximum measured plasma concentration over the time span specified
pharmacokinetic changes of niclosamide from baseline in each dose group: Tmax | follow-up 48 days after dosing
  Time of the maximum measured plasma concentration
pharmcodynamic analysis of niclosamide from baseline in each dose group and time point: CRP | on Day 3, 7, 10 and 14
  Change in C reactive protein levels

IPD SHARING:
Plan to Share IPD: No